CLINICAL TRIAL: NCT00816153
Title: Is Pleth Variability Index Able to Guide Fluid Management During Surgery?
Brief Title: Pleth Variability Index and Fluid Management During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Forget Patrice, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008/1
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Fluid Management
Keywords: Pleth variability Index; Fluid management; Fluid management during surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVI (Experimental): PVI guided fluid management
  Interventions: Other: PVI-guided fluid management
- Control (No Intervention)

INTERVENTIONS:
Other: PVI-guided fluid management — Peroperative comparison of standard care with PVI-guided fluid management (optimization of the PVI value with fluid loading)
  Arms: PVI

SUMMARY:
Pleth Variability Index (PVI) seems to be an ideal parameter to guide fluid management: dynamic parameter and non-invasive. PVI could guide fluid management during surgery and optimization of the plethysmographic-derived parameter could improve hemodynamics of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Major abdominal surgery

Exclusion Criteria:

* Refusal or inability to understand the protocol
* Arrythmia
* <18 years
* Contraindication to normal mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Hemodynamics and derived-parameters | The first 48 h

SECONDARY OUTCOMES:
All causes of morbi-mortality

CONTACTS AND LOCATIONS:
Locations (1):
- St-Luc Hospital, Brussels, Belgium